CLINICAL TRIAL: NCT00371657
Title: Obesity as a Risk Factor for Small for Gestational Age and Intrauterine Growth Restriction Infants
Brief Title: Maternal Obesity and Small for Gestational Age Infants
Status: Completed | Type: Observational
Sponsor: Oklahoma State University Center for Health Sciences (Other)
Other Study IDs: 2006017
Record Dates: First submitted 2006-08-30; First posted 2006-09-04 (Estimated); Last update posted 2008-02-04 (Estimated); Status verified 2008-01

CONDITIONS: Obesity; Small for Gestational Age
Keywords: obesity; small for gestation age; intrauterine growth restriction
MeSH Terms: conditions — Obesity; Fetal Growth Retardation

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
The purpose of this retrospective pilot study is to address the effect that obesity, in the absence of other comorbidities, has on birth weight. We wish to determine if obesity is a risk factor for small for gestational age (SGA) or intrauterine growth restricted (IUGR) infants in our clinic population. There have been many studies linking maternal obesity with fetal macrosomia, defined as fetal birth weight greater than 4500 grams. However, we have noted that a percentage of our obese patient population has delivered either an SGA or IUGR infant. SGA refers to a constitutionally small infant weighing less than the 10th percentile for age. This refers to a genetically normal infant. IUGR refers to a fetus whose growth has been restricted by influences other than normal genetics.

Our study population will consist of all women over the age 18 who delivered a term infant either by vaginal delivery or cesarean section at Tulsa Regional Medical Center between July 1st 2004 and December 31st 2005.

The diagnosis of obesity will be based upon a Body Mass Index (weight in kilograms/height in meters squared) of thirty or greater. We will look at the infant birth weight as recorded in the patient's chart. We will define SGA or IUGR as birth weight less than the 10th percentile for gestational age as defined previously. The control group will consist of women meeting the same criteria except they will have a BMI less than thirty but greater than 19.8 as low maternal weight is also a risk factor for IUGR. We will compare the average birth weight and the rates of SGA/IUGR infants between the two groups and analyze using the chi-squared method of analysis.

DETAILED DESCRIPTION:
The purpose of this retrospective pilot study is to address the effect that obesity, in the absence of other comorbidities, has on birth weight. We wish to determine if obesity is a risk factor for small for gestational age (SGA) or intrauterine growth restricted (IUGR) infants in our clinic population. There have been many studies linking maternal obesity with fetal macrosomia, defined as fetal birth weight greater than 4500 grams. However, we have noted that a percentage of our obese patient population has delivered either an SGA or IUGR infant. SGA refers to a constitutionally small infant weighing less than the 10th percentile for age. This refers to a genetically normal infant. IUGR refers to a fetus whose growth has been restricted by influences other than normal genetics. Obesity is defined as a body mass index (BMI) greater than 30 by the World Health Organization and the National Institutes of Health. This is a relevant topic in health care today as one-third of adult women fall into the category of obese. As this number increases, we will be faced with the challenge to provide comprehensive prenatal care to these women. Risk factors for IUGR in particular include hypertension, renal disease, restrictive lung disease, diabetes, cyanotic heart disease, antiphospholipid syndrome, collagen vascular disease, hemoglobinopathies, tobacco and drug use, severe malnutrition, placental disease, multiple gestation, infection, genetic disorders, and teratogenic exposure. The children born with this condition are at greater risk for hypothermia, hypoglycemia, apneic episodes, seizures, sepsis, and neonatal death. Long term problems usually develop based on the cause of the SGA or IUGR status with most catching up growth-wise to other children their age. Previous studies have linked these conditions to higher incidence of hypertension and cardiovascular problems. The most basic screening for these conditions is the simple fundal height measurement, as the most likely physical finding will be uterine size less than dates. It is questionable how accurate this measurement is in the obese population as the measurement is taken over the layer of abdominal fat. Obesity in the pregnant patient is linked to increased rates of hypertension, preeclampsia, and gestational or preexisting diabetes. Although many studies have also linked fetal macrosomia to maternal obesity, there have been studies published within the last year that relate maternal obesity with SGA or IUGR infants. A Danish study looked at a cohort of women who delivered singleton infants. They looked at pregnancy complications including diabetes, hypertension, preeclampsia, and cesarean delivery. The study population included only deliveries from 37-42 weeks gestation. Women with hypertension and preexisting diabetes were included in the study population. The findings included higher risk of macrosomic infants in the general study population. In a small segment of the study population, however, they found increased incidence of SGA infants but not IUGR infants. This hints at a possible relationship between obesity and SGA but does not control for other variables. A study out of Medical University of South Carolina looked at prepregnancy weights and subsequent weight gain. It was a cohort study using birth certificate information linked to the South Carolina Pregnancy Risk Assessment Monitoring System, a system of telephone and mail survey, to collect the data for this study. The results included a 1.8 times greater likelihood of an obese woman delivering a very low birth weight infant (3).

Study Population Inclusion/Exclusion Criteria Our study population will consist of all women over the age 18 who delivered a term infant either by vaginal delivery or cesarean section at Tulsa Regional Medical Center between July 1st 2004 and December 31st 2005. We choose this time frame as we feel this will give an adequate sample size of approximately about 160 women in the study group and about 260 in the control group, while allowing for completion of the project within 12 to 18 months. Our statistician, Dr. Mark Payton, has completed a power analysis for these numbers, and it is included with our submission. We will define a term infant as 37 weeks gestation or greater. They must have had at least one visit at the Houston Park Ob-Gyn clinic, not including the initial prenatal lab visit, before delivery. Our study population will consist of mainly Medicaid patients, most of who are of lower socioeconomic status. The ethnic blend of our study population will include Caucasian, African-American, Hispanic, American Indian, and Asian women. Our study population will have a BMI greater than or equal to 30 based on initial recorded weight and recorded height. We will exclude women with multiple gestation, hypothyroidism, hyperthyroidism, heart disease, tobacco or drug use, gestational or preexisting diabetes, autoimmune disease of any form, hypertension, collagen vascular disease, any disease process resulting in decreased gastrointestinal nutrient absorption, or lung disease as these are conditions known to be risk factors for IUGR (5).

Early Termination Criteria N/A

Methods/Procedures Diagnosis The diagnosis of obesity will be based upon initial weight and height recorded in the patients chart, typically during the first trimester, to derive a BMI (weight in kilograms/height in meters squared). Although total weight gain during a term pregnancy could add enough to the BMI to falsely indicate obesity, since we will be using the initial weight recorded, this difficulty should be minimized. The cutoff for our study group will be a BMI of thirty or greater as this is the definition of obesity by the World Health Organization and the National Institutes of Health. We will look at the infant birth weight as recorded in the patient's chart. We will define SGA or IUGR as birth weight less than the 10th percentile for gestational age as defined previously. The control group will consist of women meeting the same criteria except they will have a BMI less than thirty but greater than 19.8 as low maternal weight is also a risk factor for IUGR.

Data Collection The collaborating investigators and research assistants will collect only the following information from the patients chart: age, height, weight at initial visit, date of delivery, infant birth weight, smoking status, and any of the abovementioned comorbidities that would exclude the patient from the study. No other data will be collected from any patients chart. We will utilize research assistants in the collection of this data, and these research assistants will be OSU medical students employed by the work study program to work on this project. They will be collecting data from clinic records. They have basic human research and HIPAA training and are allowed access to patient chart information as they fall under the OSU community of individuals with this privilege. Analysis We will compare the average birth weight and the rates of SGA/IUGR infants between the two groups. We will analyze the results using chi-squared method of analysis.

Confidentiality The clinic records to be reviewed will be kept in the Houston Park medical records department which is either locked or under security supervision at all times. The hospital records will be kept in the Tulsa Regional Medical Center health information management department. This department is locked 24 hours a day. No identifying information from any individual's chart will be recorded, so de-identification will occur when the data is collected, and no master list of patient names or other identifying information will be kept.

ELIGIBILITY:
Inclusion Criteria:

* Our study population will consist of all women over the age 18 who delivered a term infant either by vaginal delivery or cesarean section at Tulsa Regional Medical Center between July 1st 2004 and December 31st 2005. They must have had at least one visit at the Houston Park Ob-Gyn clinic, not including the initial prenatal lab visit, before delivery.

Exclusion Criteria:

* We will exclude women with multiple gestation, hypothyroidism, hyperthyroidism, heart disease, tobacco or drug use, gestational or preexisting diabetes, autoimmune disease of any form, hypertension, collagen vascular disease, any disease process resulting in decreased gastrointestinal nutrient absorption, or lung disease as these are conditions known to be risk factors for IUGR.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 420
Dates: Start 2006-07; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly A. Sorensen, D.O., Principal Investigator — Oklahoma State University Center for Health Sciences
Locations (1):
- Oklahoma State University Center for Health Sciences Houston Parke Clinic, Tulsa, Oklahoma, United States

REFERENCES:
- [Background] Hulsey TC, Neal D, Bondo SC, Hulsey T, Newman R. Maternal prepregnant body mass index and weight gain related to low birth weight in South Carolina. South Med J. 2005 Apr;98(4):411-5. doi: 10.1097/01.SMJ.0000145283.69631.FC. PMID 15898514